CLINICAL TRIAL: NCT04016337
Title: Evaluación Del Efecto de Bebidas Ricas en Compuestos Bioactivos Para Modular el Metabolismo Energético en Adultos Con Sobrepeso
Brief Title: Evaluation of New Beverages Rich in Bioactive Compounds for the Modulation of Energetic Metabolism in Overweight Adults
Acronym: BEBESANO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Católica San Antonio de Murcia (Other)
Collaborators: National Research Council, Spain (Other Government)
Responsible Party: Principal Investigator, Débora Villaño, Associate Professor, Universidad Católica San Antonio de Murcia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: AGL2016-75332-C2-2-R
Record Dates: First submitted 2019-07-02; First posted 2019-07-11 (Actual); Last update posted 2019-07-19 (Actual); Status verified 2019-07

CONDITIONS: Obesity; Inflammation; Insulin Sensitivity
Keywords: sweeteners; stevia; sucralose; polyphenols; maqui; bioavailability; inflammation; gut hormones; biomarkers
MeSH Terms: conditions — Obesity; Inflammation; Insulin Resistance | interventions — Beverages

STUDY DESIGN:
Intervention Model Description: The chronic study consisted on a 60 days consumption of a beverage (330 mL) made with lemon and maqui and added a particular sweetener.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Beverages were provided by manufacturer with codes and no one, up to now, knows the sweetener added on each type.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intervention with beverage added with sucralose (Experimental): A beverage (330 mL) made with lemon and maqui extracts and sweetened with sucralose was taken by participants, during 60 days. Beverages were made in a semi-industrial process in a pilot plant. Microbiological tests, quality controls and shelf-life assays were performed following legislation on beverages.
  Concentrations of lemon and maqui extract are under industrial secret. The sweetener sucralose was added within the ranges established by law as maximums.
  The beverage was carried out in the pilot plant of a company (Nutracitrus) with all the safety systems, tested by an external lab (Ecosur), apart from the routine controls themselves.
  All ingredients were suitable for consumption and purchased from different companies with their respective certificates and conservation was at 5 º C for a maximum of 7 days, prior to administration to volunteers.
  Interventions: Dietary Supplement: Beverages
- Intervention with beverage added with saccharose (Experimental): A beverage (330 mL) made with lemon and maqui extracts and sweetened with saccharose was taken by participants, during 60 days. Beverages were made in a semi-industrial process in a pilot plant. Microbiological tests, quality controls and shelf-life assays were performed following legislation on beverages.
  Concentrations of lemon and maqui extract are under industrial secret. The sweetener saccharose was added within the ranges established by law as maximums.
  The beverage was carried out in the pilot plant of a company (Nutracitrus) with all the safety systems, tested by an external lab (Ecosur), apart from the routine controls themselves.
  All ingredients were suitable for consumption and purchased from different companies with their respective certificates and conservation was at 5 º C for a maximum of 7 days, prior to administration to volunteers.
  Interventions: Dietary Supplement: Beverages
- Intervention with beverage added with stevia (Experimental): A beverage (330 mL) made with lemon and maqui extracts and sweetened with stevia extract was taken by participants, during 60 days. Beverages were made in a semi-industrial process in a pilot plant. Microbiological tests, quality controls and shelf-life assays were performed following legislation on beverages.
  Concentrations of lemon and maqui extract are under industrial secret. The sweetener stevia was added within the ranges established by law as maximums.
  The beverage was carried out in the pilot plant of a company (Nutracitrus) with all the safety systems, tested by an external lab (Ecosur), apart from the routine controls themselves.
  All ingredients were suitable for consumption and purchased from different companies with their respective certificates and conservation was at 5 º C for a maximum of 7 days, prior to administration to volunteers.
  Interventions: Dietary Supplement: Beverages

INTERVENTIONS:
Dietary Supplement: Beverages — The beverages were all made with lemon and maqui extracts, and different sweeteners

SUMMARY:
During last decades, an excessive intake of sugars has been observed in westernized countries, mainly due to the consumption of sugar-rich soft drinks. Epidemiological studies have pointed out a positive correlation between the consumption of such drinks and the risk of obesity, diabetes, and cardiovascular diseases. Therefore, there is a growing trend looking for new non-caloric alternatives (sweeteners) in order to reduce the sugar content of foodstuffs without losing their sweetness and tastefulness. However, some questions regarding sweeteners have recently arisen as their effects after long-term consumption have not been fully unravelled. They could also contribute to a higher caloric intake and to disrupt the gut microbiota. Besides seeking new alternatives for the high intake of sugar-rich drinks, there is a need for increasing the consumption of fruits and vegetables among general public. Developing new products to stretch the shelf-life of fresh fruits, preserving their nutrients, and reducing the energetic content of fruit juices should also be accomplished. In this sense, lemon juice has been proposed as an interesting ingredient in the elaboration of soft drinks due to its distinctive aroma and high nutritive value. Its combination with maqui berry juices contributes to stabilize the colour and phenolic compounds that both products contain (mainly flavanones for lemon juice and anthocyanins for maqui). The beneficial effects of these vegetal foodstuffs and their phenolic substances on glucose intolerance have been reported.The aim of BEBESANO is studying the beneficial effects of sugar-free, rich-in-phytochemicals drink consumption on postprandial hyperglycaemia, in order to provide alternatives to excessive sugar intake and counteract the postprandial response linked to sugar consumption in subjects with low levels of chronic inflammation such as overweight people. Moreover, BEBESANO will shed light on the interactions of food constituents with the main pathways involved in the lipid and glucose metabolism, oxidative stress, inflammation, and hormonal regulation in overweight population.

DETAILED DESCRIPTION:
The effect of the consumption of fruit-based drinks, sweetened and rich in bioactive compounds has been evaluated in acute and chronic clinical studies. They have been carried out at the Catholic University of Murcia, in accordance with the Helsinki Declaration of Human Studies and approved by the official Ethical Committee of Clinical Studies (CEIC).

All participants were informed on the characteristics of the study and they signed the written-informed consent. Dietetic and life style habits were recorded from all participants. There were no drop-outs during the whole period of the study and no adverse effects were reported. Safety clinical parameters (hepatic enzymes, renal function) were measured as well.

Acute study The acute study has determined markers of intake such as metabolites generated from ingested polyphenolic compounds, as well as markers of effect, such as markers of inflammatory processes, oxidative stress, glycemic and lipid homeostasis and hormones. Specifically, the analysis of incretines in plasma using LC-MS techniques has been included.

A double-blind, randomized, cross-over clinical study has been conducted in a population of 20 overweight individuals. After an initial phase of 3 days of wash-out with a strict diet free of polyphenols and added sugars, 330 mL of the problem drink was administered on fasting conditions:

* Drink made with lemon and maqui and sweetened with saccharose
* Drink made with lemon and maqui and sweetened with sucralose
* Drink made with lemon and maqui and sweetened with stevia

Blood samples were then taken at various times (0, 15, 30, 60, 90, 120, 210 minutes). Urine samples were collected 24 hours earlier (0 point) as well as in 0-4, 4-8, 8-12, 12-24 h tranches.

After 7 days, the process was repeated again, for each volunteer to take another drink, until all the drinks were consumed by all the volunteers.

Chronic study Prolonged consumption of beverages over several weeks will allow the later modification markers, such as parameters related to inflammation or oxidative status and long-term hormonal response, to be evaluated.

The trial is randomized, double-blind, parallel, with 3 groups of 46 subjects each. The groups were randomized stratified by sex, BMI, and age. Recruitment has taken place at various Health Centers and at UCAM. Those who are able to participate have been informed of the study and asked to sign informed consent.

The study includes beverages already studied in acute intervention:

* Drink made with lemon and maqui and sweetened with saccharose
* Drink made with lemon and maqui and sweetened with sucralose
* Drink made with lemon and maqui and sweetened with stevia

Participants were advised not to change their dietary habits during the study period.

Each individual was given a type of drink (330 mL/day) for 60 days. Blood samples were taken, as well as 24h-urine, at day 0 and at the end of the study (60 days), to perform the various assessments.

ELIGIBILITY:
Inclusion Criteria:

* healthy volunteers,
* body mass index (BMI) between 25 - 29.9 kg/m2 (overweight according to WHO criteria)
* 35-55 years,
* absence of disease.

Exclusion Criteria:

* Hypertension
* Dislipemia
* Smoking

Ages: 35 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 138 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2018-03-30 (Actual); Study Completion 2018-08-31 (Actual)

PRIMARY OUTCOMES:
Changes in markers of inflammation (cytokines) | Changes observed from baseline at day 0 compared to 60 days
  Plasma levels of IL-6, TNF-alfa, IL-10
Changes in markers of inflammation (c-reactive protein) | Changes observed from baseline at day 0 compared to 60 days
  Plasma levels of c-reactive protein (mg/dL)
Changes in markers of lipid metabolism | Changes observed from baseline at day 0 compared to 60 days
  Plasma concentrations of Total cholesterol, LDL, HDL, Triglycerides
Changes in markers of glycemic metabolism | Changes observed from baseline at day 0 compared to 60 days
  Plasma levels of insulin and glucose
Insulin resistance | Changes observed from baseline at day 0 compared to 60 days
  Insulin and glucose levels will be combined to report HOMA index
Changes in hormone response | Changes observed from baseline at day 0 compared to 60 days
  Plasma levels of leptin, ghrelin
Changes in anthropometric parameters | Changes observed from baseline at day 0 compared to 60 days
  weight and height will be combined to report BMI in kg/m^2

CONTACTS AND LOCATIONS:
Overall Officials: Débora Villaño Valencia, PhD, Principal Investigator — Universidad Católica de Murcia (UCAM)
Locations (1):
- Universidad Católica de Murcia (UCAM), Guadalupe, Murcia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Villano D, Zafrilla P, Garcia-Viguera C, Dominguez-Perles R. A UHPLC/MS/MS method for the analysis of active and inactive forms of GLP-1 and GIP incretins in human plasma. Talanta. 2022 Jan 1;236:122806. doi: 10.1016/j.talanta.2021.122806. Epub 2021 Aug 19. PMID 34635208